CLINICAL TRIAL: NCT00612157
Title: Prospective, Randomized, Double-Blind, Placebo-Controlled Trial Assessing the Effect of Eszoplicone on Initial Continuous Positive Airway Pressure (CPAP) Compliance
Brief Title: Continuous Positive Airway Pressure (CPAP) Promotion And Prognosis - the Army Sleep Apnea Program (ASAP)
Acronym: CPAPASAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Christopher J. Lettieri, MD / Pulmonary, Critical Care & Sleep Medicine, Walter Reed Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: WRAMC07-17022
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Last update posted 2009-02-26 (Estimated); Status verified 2009-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Continuous Positive Airway Pressure; CPAP Compliance; Non-benzodiazepine hypnotics
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OSA CPAP (Active Comparator)
  Interventions: Drug: Eszopiclone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo control

INTERVENTIONS:
Drug: Eszopiclone — Eszopiclone 3mg orally at bedtime for 14 nights
  Other Names: Lunesta
  Arms: OSA CPAP
Drug: Placebo control — Matching placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of Eszopiclone in improving short and intermediate-term compliance with continuous positive airway pressure (CPAP) in patients newly diagnosed with obstructive sleep apnea (OSA).

DETAILED DESCRIPTION:
CPAP is the treatment of choice for patients with OSA. However, patients are frequently intolerant of this therapy initially. After continued use, tolerance is achieved. However, this initial discomfort or intolerance frequently leads to a patient-initiated discontinuation of therapy. It has been shown that CPAP use at 1 month predicts use at 6 months and 1 year. Patients who initially struggle with or are intolerant of CPAP frequently abandon therapy and are unlikely to use it long term. To prevent this, sleep physicians often prescribe short courses of sedatives to help improve initial tolerance and promote better compliance with therapy. However, the effectiveness of this practice has not been validated in a clinical trial. Compliance, in reference to this study is the willingness of the patients to follow the prescribed course of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Newly diagnosed with OSA who are prescribed CPAP therapy

Exclusion Criteria:

* Patients < 18 years old
* Patients over 65 years
* Pregnant women
* Patients with chronic liver disease
* Patients who abuse alcohol
* Patients taking narcotics or using sedative-hypnotic agents such as Ambien, Klonopin or Benadryl

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 154 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Short term CPAP Compliance | 3 months
Intermediate CPAP Compliance | 1 year

SECONDARY OUTCOMES:
Quality of Life Issue - Prostate Symptoms for men | 1 month, 3 months, 6 months, 9 months, 12 months
Quality of Life Issue - Erectile Dysfunction for men | 1 month, 3 months, 6 months, 9 months, 12 months
Quality of Life Issue - Sleepiness | 1 month, 3 months, 6 months, 9 months, 12 months
Quality of Life Issue - Fatigue | 1 month, 3 months, 6 months, 9 months, 12 months
Quality of Life Issue - Subjective Sleep Quality | 1 month, 3 months, 6 months, 9 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Lettieri, MD, Principal Investigator — Walter Reed Army Medical Center
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Lettieri CJ, Eliasson AH, Andrada T, Khramtsov A, Raphaelson M, Kristo DA. Obstructive sleep apnea syndrome: are we missing an at-risk population? J Clin Sleep Med. 2005 Oct 15;1(4):381-5. PMID 17564406
- [Background] Quera-Salva MA, McCann C, Boudet J, Frisk M, Borderies P, Meyer P. Effects of zolpidem on sleep architecture, night time ventilation, daytime vigilance and performance in heavy snorers. Br J Clin Pharmacol. 1994 Jun;37(6):539-43. doi: 10.1111/j.1365-2125.1994.tb04301.x. PMID 7917771
- [Background] Feinberg I, Maloney T, Campbell IG. Effects of hypnotics on the sleep EEG of healthy young adults: new data and psychopharmacologic implications. J Psychiatr Res. 2000 Nov-Dec;34(6):423-38. doi: 10.1016/s0022-3956(00)00038-8. PMID 11165310
- [Background] Blois R, Gaillard JM, Attali P, Coquelin JP. Effect of zolpidem on sleep in healthy subjects: a placebo-controlled trial with polysomnographic recordings. Clin Ther. 1993 Sep-Oct;15(5):797-809. PMID 8269446
- [Background] Ballester E, Badia JR, Hernandez L, Carrasco E, de Pablo J, Fornas C, Rodriguez-Roisin R, Montserrat JM. Evidence of the effectiveness of continuous positive airway pressure in the treatment of sleep apnea/hypopnea syndrome. Am J Respir Crit Care Med. 1999 Feb;159(2):495-501. doi: 10.1164/ajrccm.159.2.9804061. PMID 9927363
- [Derived] Lettieri CJ, Shah AA, Holley AB, Kelly WF, Chang AS, Roop SA; CPAP Promotion and Prognosis-The Army Sleep Apnea Program Trial. Effects of a short course of eszopiclone on continuous positive airway pressure adherence: a randomized trial. Ann Intern Med. 2009 Nov 17;151(10):696-702. doi: 10.7326/0003-4819-151-10-200911170-00006. PMID 19920270